CLINICAL TRIAL: NCT02579252
Title: A 24 Months Randomised, Placebo-controlled, Parallel Group, Double Blinded, Multi Centre, Phase 2 Study to Assess Safety and Efficacy of AADvac1 Applied to Patients With Mild Alzheimer's Disease
Brief Title: 24 Months Safety and Efficacy Study of AADvac1 in Patients With Mild Alzheimer's Disease
Acronym: ADAMANT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axon Neuroscience SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-AD-003; 2015-000630-30 (EudraCT Number)
Record Dates: First submitted 2015-10-09; First posted 2015-10-19 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Alzheimer's Disease
Keywords: vaccine; tau protein; active; immunization; KLH; immunotherapy; tau
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia; Motor Activity; Pick Disease of the Brain | interventions — AADvac1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AADvac1 (Experimental): AADvac1 is a suspension for subcutaneous injection. AADvac1 is provided in single-use vials. Dosage: 40 µg Axon peptide 108 (coupled to keyhole limpet haemocyanin (KLH)) using aluminium hydroxide (containing 0.5 mg Al3+) as adjuvant, in a phosphate buffer.
  Patients receive 6 doses in 4-week intervals, and then 5 individual booster doses in 3-month intervals, for a total of 11 doses.
  Interventions: Biological: AADvac1
- Placebo (Placebo Comparator): Placebo is a suspension for subcutaneous injection. Placebo is provided in single-use vials. Dosage: aluminium hydroxide (containing 0.5 mg Al3+), in a phosphate buffer. Patients receive 6 doses in 4-week intervals, and then 5 individual booster doses in 3-month intervals, for a total of 11 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AADvac1
  Arms: AADvac1
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the safety and efficacy of AADvac1 in the treatment of patients with mild Alzheimer's disease.

60% of participants will receive AADvac1 and 40% of participants will receive placebo.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a chronic progressive neurodegenerative disorder of the brain. Over the course of the disease, pathological proteins accumulate in the brain, damaging neurons, thus causing them to lose their connections and die.

Currently available treatments are designed to compensate for the neurotransmitter loss caused by the disease without affecting the disease process itself.

AADvac1 is designed to raise antibodies against pathological tau protein (the primary constituent of neurofibrillary pathology in AD). These antibodies are expected to prevent tau protein from aggregating, to facilitate the removal of tau protein aggregates and prevent the spreading of pathology, slowing or halting the progress of the disease.

ELIGIBILITY:
Inclusion criteria (abbreviated):

* Diagnosis of probable Alzheimer's disease according to the revised National Institute on Aging-Alzheimer's Association (NIA-AA) criteria (McKhann 2011).
* Mini Mental State Examination (MMSE) score ≥ 20 and ≤ 26.
* Brain MRI finding consistent with the diagnosis of Alzheimer's disease
* Medial temporal lobe atrophy: Scheltens score of ≥ 2 (on a scale of 0-4 on the more atrophied side) AND/OR positive AD biomarker profile in the CSF (amyloid+, tau+)
* At least 6 years of formal elementary education.
* Age 50-85 years.
* Fluency in the local language and sufficient auditory and visual capacities to allow neuropsychological testing.
* Ability to read and understand the informed consent.
* Stable therapy with an acetylcholinesterase inhibitor for at least 3 months prior to screening.
* If the patient is on memantine treatment, the dose regimen must be stable for at least 3 months prior to screening.
* Hachinski Ischemia Scale score ≤ 4.
* Availability of a caregiver.
* Female patients must be either surgically sterile or at least 2 years postmenopausal.
* Male patients must either be surgically sterile, or he and his female spouse/partner who is of childbearing potential must be using highly effective contraception starting at screening and continuing throughout the study period.
* Patient provides written informed consent.

Exclusion criteria (abbreviated):

* Participation in another clinical study within 3 months prior to screening.
* Pregnant or breastfeeding female.
* Not expected to complete the clinical study.
* Known allergy to components of the vaccine.
* Contraindication for MRI imaging.
* Any of the following detected by brain MRI:

  * Infarction in the territory of large vessels
  * More than one lacunar infarct.
  * Any lacunar infarct in a strategically important location.
  * Confluent hemispheric deep white matter lesions (Fazekas grade 3).
  * Other focal lesions which may be responsible for the cognitive status of the patient or any other abnormalities associated with significant central nervous disease other than Alzheimer's disease.
* Surgery (under general anaesthesia) within 3 months prior to screening and/or scheduled surgery (under general anaesthesia) during the whole study period.
* Patient has a history and/or currently suffers from a clinically significant autoimmune disease, or is expected to receive immunosuppressive or immunomodulatory treatment at the present or in the future.
* Recent history of cancer (last specific treatment ≤ 5 years prior to Screening).
* Myocardial infarction within 2 years prior to screening.
* Hepatitis B, C, HIV or Syphilis.
* Active infectious disease.
* Presence and/or history of immunodeficiency.
* Patient currently suffering from a clinically important systemic illness:

  * poorly controlled congestive heart failure (NYHA ≥ 3)
  * BMI > 40
  * poorly controlled diabetes (HbA1c > 7.5%)
  * severe renal insufficiency (eGFR < 30 mL/min)
  * chronic liver disease - ALT (alanine aminotransferase) > 66 U/L in females or > 80 U/L in males, AST (aspartate aminotransferase) > 82 U/L
  * QTc interval prolongation in ECG (> 450 ms)
  * other clinically significant systemic illness, if considered relevant by the investigator
* Hypothyroidism, defined as TSH (thyroid-stimulating hormone) elevation > 5.000 mcIU/mL, and/or FT4 levels < 0.7 ng/dL. Patients with corrected hypothyroidism are eligible for the study provided that treatment has been stable for 3 months before study entry.
* Valid diagnosis of a significant psychiatric illness such as schizophrenia, any type of psychotic disorder or bipolar affective disorder.
* Current depressive episode (Geriatric Depression Scale GDS ≥ 6) or major depressive episode within the last 1 years.
* Metabolic or toxic encephalopathy or dementia due to a general medical condition.
* History of alcohol or drug abuse or dependence within the past 2 years.
* Wernicke's encephalopathy.
* History or evidence of any CNS disorder other than AD that could be the cause of dementia.
* Cerebrovascular disease (ischemic or haemorrhagic stroke), or diagnosis of possible, probable or definite vascular dementia.
* Epilepsy.
* Treatment with experimental immunotherapeutics including intravenous immunoglobulin within 3 months prior to screening.
* Treatment with experimental therapies for AD aiming at disease-modification within 3 months prior to screening.
* Patient is currently being treated or was treated in the past with any active vaccines for AD.
* Treatment with immunosuppressive drugs.
* Change in dose of previous and current medications within the last 30 days prior to Screening (V01), if considered clinically relevant by the investigator.
* Vitamin B12 deficiency (serum vitamin B12 < 191 pg/mL).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2016-03; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Safety (all-case treatment-emergent adverse events except local reactions) | 24 months
  The safety and tolerability of AADvac1 in the treatment of patients with mild Alzheimer disease, as assessed by AEs, vital signs, ECG, laboratory measures, MRI of the brain, physical and neurological examination, Columbia Suicide Severity Rating Scale (C-SSRS) and review of the Patient Diary

SECONDARY OUTCOMES:
Clinical Dementia Rating (CDR) Sum of Boxes | 24 months
  The domain scores of the standard 6-domain CDR assessment will be summed up to obtain a Sum-of-Boxes score of 0-18
Custom cognitive battery (composite standard score) | 24 months
  A composite standard score will be calculated from the following tests:
  Cogstate International Shopping List Task (memory)
  * immediate free recall
  * delayed free recall
  * delayed recognition
  Cogstate One Card Learning Task (memory)
  Cogstate One Card Back Task (memory)
  Category Fluency Test (executive function, language)
  Letter Fluency Test (executive function, language)
  Digit Symbol Coding (executive functioning, working memory and processing speed)
Alzheimer's Disease Cooperative Study - Activities of Daily Living questionnaire (version for Mild Cognitive Impairment) (ADCS MCI ADL) | 24 months
  Activities of daily living will be assessed using the informant-based ADCS questionnaire (both the score for the 18-point and the 24-point version will be calculated)
Immunogenicity | 24 months

OTHER OUTCOMES:
Exploratory: Fludeoxyglucose Positron Emission Tomography (FDG PET) assessment of brain metabolism (change in cerebral glucose metabolic rate expressed as Standardised Uptake Value Ratio [SUVR] change, multiple regions of interest) | 24 months
Exploratory: MRI volumetry | 24 months
Exploratory: Cerebrospinal fluid (CSF) biomarkers | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Schmidt, Prof. MD., Principal Investigator — Medical University, Graz, Austria
Locations (42):
- Austria (4):
  - Ordination Dr. Bancher, Horn, Lower Austria
  - Universitätsklinik für Neurologie, Graz, Styria
  - Abteilung Psychiatrie und Psychotherapie, LKH Hall, Hall in Tirol, Tyrol
  - Universitätsklinikum Innsbruck, Innsbruck, Tyrol
- Czechia (5):
  - Fakultni nemocnice u sv. Anny v Brne, Mezinarodni centrum klinickeho vyzkumu (ICRC), Centrum pro kognitivni poruchy, Neuro 2, Brno
  - Fakultni nemocnice Hradec Kralove, Neurologicka Klinika, Hradec Králové
  - Narodni ustav dusevniho zdravi (NÚDZ), Department of cognitive disorders - AD Center, Klecany
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
- Germany (6):
  - Neuro Centrum Odenwald, Erbach, Rhineland-Palatinate
  - Arzneimittelforschung Leipzig (AFL), Leipzig, Saxony
  - Universität Heidelberg, Zentralinstitut für Seelische Gesundheit, Mannheim
  - Klinikum rechts der Isar der Technischen Universität München, Klinik und Poliklinik fur Psychiatrie und Psychotherapie, München
  - Praxis Dr. Klaus Christian Steinwachs, Nuremberg
  - Universitätsklinikum Ulm, Klinik und Poliklinik für Neurologie, Ulm
- Poland (11):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - Pallmed prowadzacy NZOZ Dom Sue Ryder w Bydgoszczy Centrum Psychoneurologii Wieku Podeszlego, Bydgoszcz
  - Wielospecjalistyczna Poradnia Lekarska Synapsis, Katowice
  - Care Clinic, Katowice
  - Centrum Neurologii Klinicznej, Krakowska Akademia Neurologii, Krakow
  - KO-MED Centra Kliniczne Sp. z o.o., Lublin
  - Oddzial Neurologiczny, Olsztyn
  - NZOZ Neuro-Kard, Poznan
  - EUROMEDIS Sp. z o.o., Szczecin
  - Centrum Medyczne NeuroProtect, Warsaw
  - Wrocławskie Centrum Alzheimerowskie, Wroclaw
- "Dr. Constantin Gorgos" Psychiatry Hospital Titan, Bucharest, Romania
- Slovakia (9):
  - Neurologicka ambulancia, Banská Bystrica
  - Nestatna psychiatricka ambulancia, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica Stare Mesto, I. Neurologicka klinika LF UK a UNB, Bratislava
  - Univerzitna nemocnica Bratislava, Psychiatricka klinika LFUK a UNB, Bratislava
  - Univerzitna nemocnica L Pasteura Kosice, Psychiatricka klinika, Košice
  - NEURES, s.r.o. Neurologicka ambulancia, Krompachy
  - Centrum zdravia R.B.K., s.r.o., Psychiatricka ambulancia, Svidník
  - Pro Mente Sana S.R.O., Psychiatricka Ambulancia, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina, Psychiatricke oddelenie, Žilina
- Slovenia (2):
  - Univerzitetni klinični Center Ljubljana, Neurology Clinic, Ljubljana
  - University Clinical Centre Maribor, Maribor
- Sweden (4):
  - Skånes Universitetssjukhus Malmö, Minneskliniken, Malmo
  - Sahlgrenska Universitetssjukhuset, Minnesmottagningen, Mölndal
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Akademiska Sjukhuset I Uppsala, Minnes-och geriatrikmottagningen, Uppsala

REFERENCES:
- [Background] Kontsekova E, Zilka N, Kovacech B, Skrabana R, Novak M. Identification of structural determinants on tau protein essential for its pathological function: novel therapeutic target for tau immunotherapy in Alzheimer's disease. Alzheimers Res Ther. 2014 Aug 1;6(4):45. doi: 10.1186/alzrt277. eCollection 2014. PMID 25478018
- [Background] Kontsekova E, Zilka N, Kovacech B, Novak P, Novak M. First-in-man tau vaccine targeting structural determinants essential for pathological tau-tau interaction reduces tau oligomerisation and neurofibrillary degeneration in an Alzheimer's disease model. Alzheimers Res Ther. 2014 Aug 1;6(4):44. doi: 10.1186/alzrt278. eCollection 2014. PMID 25478017
- [Background] Novak P, Schmidt R, Kontsekova E, Zilka N, Kovacech B, Skrabana R, Vince-Kazmerova Z, Katina S, Fialova L, Prcina M, Parrak V, Dal-Bianco P, Brunner M, Staffen W, Rainer M, Ondrus M, Ropele S, Smisek M, Sivak R, Winblad B, Novak M. Safety and immunogenicity of the tau vaccine AADvac1 in patients with Alzheimer's disease: a randomised, double-blind, placebo-controlled, phase 1 trial. Lancet Neurol. 2017 Feb;16(2):123-134. doi: 10.1016/S1474-4422(16)30331-3. Epub 2016 Dec 10. PMID 27955995
- [Derived] Kovacech B, Cullen NC, Novak P, Hanes J, Kontsekova E, Katina S, Parrak V, Fresser M, Vanbrabant J, Feldman HH, Winblad B, Stoops E, Vanmechelen E, Zilka N. Post hoc analysis of ADAMANT, a phase 2 clinical trial of active tau immunotherapy with AADvac1 in patients with Alzheimer's disease, positive for plasma p-tau217. Alzheimers Res Ther. 2024 Nov 23;16(1):254. doi: 10.1186/s13195-024-01620-7. PMID 39580468